## Child Characteristics, Neuromarkers, and Intervention Components Impacting Treatment Outcome: CCT, TF-CBT, TAU

NCT02926677

9/18/20

Victor G. Carrion, Principal Investigator Stanford University Stanford, California 94305

Planned Sample Size: Analyses will be conducted on data for participants that completed treatment from baseline to month 3 (end of treatment). The sample size is 8 participants for the CCT group, 8 for TF-CBT, and 6 for TAU.

Planned Analyses: Factorial ANOVAs comparing baseline to month 3 (end of treatment) total scores on all outcome measures (UCLA PTSD Reaction Index for DSM 5 child and parent versions, Child Depression Inventory, Multidimensional Anxiety Scale for Children, Behavior Rating Inventory of Executive Function) will be conducted for each treatment arm.